CLINICAL TRIAL: NCT01379898
Title: Pheochromocytoma Randomised Study Comparing Adrenoreceptor Inhibiting Agents for Preoperative Treatment
Brief Title: Phenoxybenzamine Versus Doxazosin in PCC Patients
Acronym: PRESCRIPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other); UMC Utrecht (Other); VU University of Amsterdam (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Leiden University Medical Center (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); St. Antonius Hospital (Other); Medisch Spectrum Twente (Other); Maxima Medical Center (Other); Canisius-Wilhelmina Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Atrium Medical Center (Other); Isala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESCRIPT2010.369; 2010:022417-25 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-06-23 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pheochromocytoma
Keywords: Pheochromocytoma; Doxazosin; Phenoxybenzamine
MeSH Terms: conditions — Pheochromocytoma | interventions — Phenoxybenzamine; Doxazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenoxybezamine (Active Comparator): Phenoxybenzamine (capsules 10 mg, once to twice daily) is administered orally, starting 2-3 weeks before planned resection of PCC.
  Interventions: Drug: Phenoxybenzamine
- Doxazosin (Active Comparator): Phenoxybenzamine (slow release tablets 4 or 8 mg, once to twice daily) is administered orally, starting 2-3 weeks before planned resection of PCC.
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Phenoxybenzamine — Starting dosage of phenoxybenzamine in hypertensive subjects:20 mg q.d. (=10 mg b.i.d.) and in normotensive subjects 10 mg q.d. (in the evening). Dose escalation until blood pressure targets are reached, with a maximum dose of 140 mg q.d. (=70 mg b.i.d.)
  Other Names: Dibenzyran
  Arms: Phenoxybezamine
Drug: Doxazosin — Starting dosage of doxazosine in hypertensive subjects:8 mg q.d. (=4 mg b.i.d.)and in normotensive subjects starting dose 4 mg q.d. (in the evening). Dose escalation until blood pressure targets are reached, with a maximum dose of 48 mg q.d. .(=24 mg b.i.d.)
  Other Names: Cardura
  Arms: Doxazosin

SUMMARY:
* Rationale: The optimal preoperative medical management for patients with a pheochromocytoma is currently unknown. In particular, there is no agreement with respect to whether phenoxybenzamine or doxazosin is the optimal alfa-adrenoreceptor antagonist to be administered before surgical resection of a pheochromocytoma. We hypothesized that the competitive alfa1-antagonist doxazosin is superior to the non-competitive alfa1- and alfa2-antagonist phenoxybenzamine.
* Objective: comparing effects of preoperative treatment with either phenoxybenzamine or doxazosin on intraoperative hemodynamic control in patients undergoing surgical resection of a pheochromocytoma.
* Study design: Randomised controlled open-label trial.
* Study population: 18 - 55 yr old. Adult patients with a recently diagnosed benign pheochromocytoma.
* Intervention: Patients are randomised to receive oral treatment with either phenoxybenzamine or doxazosin preoperatively.
* Main study parameters/endpoints: The main study parameter is defined as the percentage of intraoperative time that blood pressure is outside the predefined target range after pretreatment with either phenoxybenzamine or doxazosin.

In this multicenter trial, we compare the effects of two commonly used drugs in patients being medically prepared for resection of a benign pheochromocytoma. Participants are not subjected to an experimental treatment of any kind, as we merely aim to describe in detail the perioperative course in general and, in particular, the intraoperative hemodynamic control in patients treated preoperatively with either phenoxybenzamine or doxazosin. A routine diagnostic work-up for pheochromocytoma will be performed in all participants. One extra blood sample (volume: 48,5 mL) is drawn before start of the study medication, and participants need to record their symptoms in a diary. In addition, patients who are pretreated in the outpatient clinic monitor their blood pressure and pulse rate at home with an automated device. Treatment with an alfa-adrenoreceptor antagonist is initiated at least 2 - 3 weeks prior to surgery. Patients who are admitted to the hospital for pretreatment with an alfa-adrenoreceptor antagonist have their blood pressure and pulse rate measured by the nursing staff. The final site visit is planned at 30 days after surgery, in line with current practice.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Pheochromocytoma (PCC) is a rare but clinically important catecholamine secreting neuro-endocrine tumour that typically arises from the adrenal gland. In addition, this neuro-endocrine tumour can also originate from chromaffin cells in sympathetic ganglia(1)(2). In this protocol, PCC refers to both adrenal and extra-adrenal chromaffin tumours with hypersecretion of catecholamines (i.e. norepinephrine and/or epinephrine). The annual incidence rate in the US population has been estimated to be 1-2 cases per 100,000 adult individuals (3). Data on the incidence and prevalence of PCC in the Netherlands have not been published. Based on the Dutch registry of pathology diagnoses (PALGA), we found an incidence of 117 cases of PCC in the year 2007 (unpublished observation).

   PCCs may occur as part of an autosomal dominant inherited tumor syndrome, caused by germline mutations in the RET proto-oncogene (Multiple Endocrine Neoplasia type 2 syndrome), VHL gene (von Hippel-Lindau disease), NF1 gene (Neurofibromatosis type 1), or in one of the genes encoding the subunits of mitochondrial complex II, also called succinate dehydrogenase (SDHB, SDHC, SDHD)(4). PCCs are termed 'sporadic' when the family history for PCC is negative. Overall, about 25% of all PCC patients harbour a germline mutation. Notably, germline mutations in one of the PCC susceptibility genes may also be present in a significant number of patients with a sporadic PCC, with mutation rates varying between 7.5 - 14.6% in the populations studied(5-7). Therefore, genetic testing is recommended in all patients with PCC(7). Very recently, a new PCC susceptibility gene has been described, and it seems likely that future research will result in the discovery of other genetic mutations associated with PCC(8).

   PCC constitutes a surgically curable cause of hypertension. Hypertension in patients with PCC can be either persistent or paroxysmal, but is absent in a minority of patients. It is a potentially life-threatening disease with a high risk for cardiovascular complications such as myocardial infarction, arrhythmias, cardiomyopathy, stroke and pulmonary edema(1). The clinical picture results from release of catecholamines by the tumour. This release can be evoked by stimuli that would normally not pose a hazard, such as surgery or general anaesthesia. Thus, preoperative treatment with alpha-adrenoceptor antagonists is usually recommended for prevention of these serious and potentially fatal complications(9). In one of the largest surgical series reported so far, perioperative mortality and morbidity were 2.4% and 23.6%, respectively(10).

   According to the literature, about 10% of the patients with PCC are normotensive(1). A normal blood pressure at diagnosis is relatively frequent among carriers of one the aforementioned germline mutations, as these individuals are subjected to periodic biochemical screening for the presence of PCC. It has been demonstrated that intraoperative hemodynamic instability during adrenalectomy for PCC occurred to the same extent in MEN2a patients (most of whom were normotensive) as in patients without MEN2a (most of whom were hypertensive)(11). Thus, preoperative treatment with alpha -adrenoceptor antagonists is also recommended for normotensive patients with PCC (9,11), Historically, the noncompetitive and nonselective alpha -adrenoceptor antagonist phenoxybenzamine has been the drug of choice(12). Alternatively, doxazosin - a competitive and selective alpha 1-adrenoceptor antagonist - might be at least as effective asphenoxybenzamine with fewer side effects. Notably, it has been suggested that doxazosin results in a significant and clinically relevant reduction of postoperative hypotension(13). Severe postoperative hypotension necessitates admission to the intensive care unit (ICU), where volume resuscitation and norepinephrine are administered under strict monitoring of hemodynamics. Data on the optimal preoperative pharmacological management of patients with PCC are conflicting. For example, a recent study reported comparable effects of phenoxybenzamine and doxazosin on intraoperative hemodynamic control(14).This study, however, was retrospective in design and therefore affected by several confounding factors such as lack of randomisation, non-standardised intraoperative care, and use of historical controls. Until now, prospective randomised controlled trials comparing phenoxybenzamine and doxazosin have not been conducted. Thus, the preoperative drug therapy of choice remains an unresolved issue, and at a recent international PCC symposium it was concluded that no specific recommendations can be made on this subject(9). We performed a survey among all university medical centers in the Netherlands, showing that almost half of the centers prescribed phenoxybenzamine, whereas the other centers used doxazosine as the preoperative drug of choice for patients with PCC(15). Usually, these drugs are administered during 2-3 weeks before surgery. This preoperative medical preparation takes place either in the outpatient or inpatient clinic, depending on patient-related factors (e.g. disease severity, geographical considerations) and local experience.

   Preoperative volume expansion is recommended in all patients with PCC(9). The rationale behind this recommendation is based on the notion that PCC is associated with a decreased intravascular volume, which is restored under influence of treatment with alpha -adrenoceptor antagonists. Without administration of volume expansion severe hypotension might ensue. Therefore, it is common practice to advise a liberal salt intake during alpha -adrenoceptor antagonist therapy and to administer a saline infusion (e.g. 2L NaCL 0.9% in 24 hours) shortly before surgery(9,15).

   Several drugs, including certain anaesthetics, may evoke an uncontrolled catecholamine release with resulting severe hemodynamic instability(16). Patients are advised to carry a document enlisting all medications which are contra-indicated in case of a PCC. There is no consensus on the optimal anaesthetic management during resection of a PCC, as randomised controlled trials on this subject are not available(16,17). In a survey on the anaesthetic management of PCC in the Netherlands, we found as many different protocols as the number of hospitals (=10) which had responded (including all university medical centers; unpublished observation).

   PRESCRIPT represents the first randomised controlled trial comparing the effects of pretreatment with either phenoxybenzamine or doxazosin on the intraoperative hemodynamic control in patients with PCC. The relevance of conducting a trial as described in this study protocol was recently expressed again by experts in the field of PCC research(18). In addition, PRESCRIPT provides a unique opportunity to prospectively collect data containing detailed information on items such as presenting symptoms and signs, perioperative outcome and results of biochemical, imaging and genetic studies in patients with PCC. Of interest, results of this study are expected to have a direct impact on national and international guidelines regarding the perioperative care of patients with PCC.
2. OBJECTIVES Primary Objective: The primary objective is to determine which of two commonly used drugs for preoperative management provides the best intraoperative hemodynamic control in patients undergoing resection of a PCC.

   Secondary Objective(s):
   * to identify other determinants of intraoperative hemodynamic control. Potential determinants are: gender or age of the patient, clinical setting for preoperative management (i.e. outpatient or inpatient clinic), preoperative levels, of catecholamines or N-terminal pro-brain-type natriuretic peptide (NT-proBNP) PCC size, sporadic or hereditary PCC,
   * to describe prospectively symptoms and signs of PCC in a large cohort of patients. Note: until now, data on symptoms and signs have been described retrospectively
   * to describe prospectively the results of several diagnostic techniques
   * to assess prospectively the distribution of sporadic and hereditary PCC in a large cohort of Dutch patients
   * to build a biobank with blood and tissue samples for future studies on PCC
3. STUDY DESIGN Randomised open-label controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diagnosis of benign Pheochromocytoma (adrenal or extra-adrenal, sporadic or hereditary:

  * hypertension
  * elevated plasma and/or urinary (nor)metanephrines. From each patient, a blood sample is collected for measurement of plasma (nor)metanephrines with the reference laboratory assay (i.e. XLC-MS/MS) at the Department of Laboratory Medicine of the UMCG.
  * localisation of PCC by anatomical (MRI/CT) and functional imaging (I123-MIBG scintigraphy or 18F-DOPA PET)
* planned for surgical removal of the PCC

Exclusion Criteria:

* age < 18 years
* malignant PCC, i.e. presence of lesions on imaging studies suggestive of distant metastases
* severe hemodynamic instability before surgery necessitating admission to intensive care unit
* pregnancy
* incapability to adhere to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-12; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The main study parameter is defined as the percentage of intraoperative time that blood pressure is outside the predefined target range after pretreatment with either phenoxybenzamine or doxazosin. | Duration of surgery, i.e. on average 3 hours
  Blood pressure and heart rate will be monitored continuesly during surgery.

SECONDARY OUTCOMES:
To attain preoperative blood pressure target values without co-medication | an expected average of 2 to 6 weeks before surgery
  success rate of doxazosin and phenoxybenzamine to attain preoperative blood pressure target values without co-medication
Resolution of (paroxysmal) symptoms and signs of pheochromocytoma. | an expected average of 2-6 weeks before surgery
  Resulution of headache, palpitations, sweeting, paleness, nausea, flushes, fatigue and anxiety.
Need for additional antihypertensive agents | an expected average of 2-6 weeks before surgery
  Assessment of the number of patients who need additional antihypertensive drugs on top of the study drugs
Adverse effects of study medication | an expected average of 2-6 weeks before surgery
  Adverse effects of doxazosin or phenoxybenzamine
Length of preoperative treatment in either outpatient or inpatient clinic. | an expected average of 2-6 weeks before surgery
  Comparing duration of preoperative treatment in either outpatient or inpatient clinic
Control of blood pressure and heart rate. | Duration of surgery, i.e. on average 3 hours
  * number of episodes with systolic blood pressure (SBP) > 160 mmHg
  * number of episodes with mean arterial blood pressure (MAP) < 60 mmHg
  * duration (in minutes) of SBP > 160 mmHg
  * duration (in minutes) of MAP < 60 mmHg
  * number of episodes with heart rate > 100/min
  * duration (in minutes) of heart rate > 100/min
  * amount and type of vasoactive agents needed during surgery for adequate blood pressure control.
  * cumulative amount and type of intravenous fluids administered
Length of hospital stay. | Participants will be followed for the duration of hospital stay an expected average of 2-5 weeks.
  Number of days the patient is staying in the hospital before and after surgery
Composite semi-quantitative score of intra- and postoperative hemodynamic control. | During surgery and the first 24 hours after surgery at the intensive/ medium care unit
  Composite semi-quantitative score of intra- and postoperative hemodynamic control based on the following parameters:
  * blood pressure and heart rate outside target range
  * need for administration of vasoactive agents
  * need for administration of intravenous fluids
Postoperative hypoglycaemia | First 24 hours postoperative
  Frequency and severity (in mmol/L)of hypoglycaemia during first 24 hours after surgery.
Perioperative mortality. | From first administration of study medication until 30 days after surgery.
  Death from any cause occurring during period from first administration of study medication until 30 days after surgery.
Perioperative cardiovascular morbidity. | From first administation of study medicaion until 30 days after surgery.
  Cardiovascular events occurring during period from first administration of study medication until 30 days after surgery. Cardiovascular events are: myocardial infarction, cardiac arrhythmia requiring medical intervention, heart failure, cerebrovascular ischemia, cerebrovascular haemorrhage.
Composite endpoint of perioperative mortality and perioperative cardiovascular morbidity. | From first administration of study medication until 30 days after surgery.
  Death from any cause occurring or cardiovascular events occurring during period from first administration of study medication until 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel N. Kerstens, MD PhD, Study Director — University Medical Center Groningen; Thera P. Links, MD PhD, Principal Investigator — University Medical Center Groningen; Gütz J. Wietasch, MD PhD, Principal Investigator — University Medical Center Groningen; Jaques W. Lenders, MD PhD, Principal Investigator — UMC St Radboud Nijmegen; G D. Valk, MD PhD, Principal Investigator — UMC Utrecht; E M. Eekhoff, MD PhD, Principal Investigator — Free University UMC Amsterdam; P H. Bisschop, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); R A Feelders, MD PhD, Principal Investigator — Erasmus Medical Center; Bas Havekes, MD PhD, Principal Investigator — Maastricht University Medical Center; Peter Oomen, MD PhD, Principal Investigator — medical center leeuwarden; I Eland, MD PhD, Principal Investigator — St. Antonius Ziekenhuis Nieuwegein; P H. Geelhoed- Duijvestijn, MD PhD, Principal Investigator — Medical Center Haaglanden; P Groote Veldman, MD PhD, Principal Investigator — Medisch Spectrum Twente; H R Haak, MD PhD, Principal Investigator — Máxima Medisch Centrum; J R. Meinardi, MD PhD, Principal Investigator — Canisius-Wilhelmina Hospital; C B. Brouwer, MD PhD, Principal Investigator — Canisius-Wilhelmina Hospital; P L. van Battum, MD, Principal Investigator — Atrium Medical Center; A A. Franken, MD PhD, Principal Investigator — Isala
Locations (1):
- Department of Endocrinology, University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Lenders JW, Eisenhofer G, Mannelli M, Pacak K. Phaeochromocytoma. Lancet. 2005 Aug 20-26;366(9486):665-75. doi: 10.1016/S0140-6736(05)67139-5. PMID 16112304
- [Background] Lenders JW, Eisenhofer G, Armando I, Keiser HR, Goldstein DS, Kopin IJ. Determination of metanephrines in plasma by liquid chromatography with electrochemical detection. Clin Chem. 1993 Jan;39(1):97-103. PMID 8419068
- [Background] Beard CM, Sheps SG, Kurland LT, Carney JA, Lie JT. Occurrence of pheochromocytoma in Rochester, Minnesota, 1950 through 1979. Mayo Clin Proc. 1983 Dec;58(12):802-4. PMID 6645626
- [Background] Neumann HP, Cybulla M, Shibata H, Oya M, Naruse M, Higashihara E, Terachi T, Ling H, Takami H, Shuin T, Murai M. New genetic causes of pheochromocytoma: current concepts and the clinical relevance. Keio J Med. 2005 Mar;54(1):15-21. doi: 10.2302/kjm.54.15. PMID 15832076
- [Background] Amar L, Bertherat J, Baudin E, Ajzenberg C, Bressac-de Paillerets B, Chabre O, Chamontin B, Delemer B, Giraud S, Murat A, Niccoli-Sire P, Richard S, Rohmer V, Sadoul JL, Strompf L, Schlumberger M, Bertagna X, Plouin PF, Jeunemaitre X, Gimenez-Roqueplo AP. Genetic testing in pheochromocytoma or functional paraganglioma. J Clin Oncol. 2005 Dec 1;23(34):8812-8. doi: 10.1200/JCO.2005.03.1484. PMID 16314641
- [Background] Korpershoek E, Van Nederveen FH, Dannenberg H, Petri BJ, Komminoth P, Perren A, Lenders JW, Verhofstad AA, De Herder WW, De Krijger RR, Dinjens WN. Genetic analyses of apparently sporadic pheochromocytomas: the Rotterdam experience. Ann N Y Acad Sci. 2006 Aug;1073:138-48. doi: 10.1196/annals.1353.014. PMID 17102080
- [Background] Gimenez-Roqueplo AP, Lehnert H, Mannelli M, Neumann H, Opocher G, Maher ER, Plouin PF; European Network for the Study of Adrenal Tumours (ENS@T) Pheochromocytoma Working Group. Phaeochromocytoma, new genes and screening strategies. Clin Endocrinol (Oxf). 2006 Dec;65(6):699-705. doi: 10.1111/j.1365-2265.2006.02714.x. PMID 17121518
- [Background] Qin Y, Yao L, King EE, Buddavarapu K, Lenci RE, Chocron ES, Lechleiter JD, Sass M, Aronin N, Schiavi F, Boaretto F, Opocher G, Toledo RA, Toledo SP, Stiles C, Aguiar RC, Dahia PL. Germline mutations in TMEM127 confer susceptibility to pheochromocytoma. Nat Genet. 2010 Mar;42(3):229-33. doi: 10.1038/ng.533. Epub 2010 Feb 14. PMID 20154675
- [Background] Pacak K, Eisenhofer G, Ahlman H, Bornstein SR, Gimenez-Roqueplo AP, Grossman AB, Kimura N, Mannelli M, McNicol AM, Tischler AS; International Symposium on Pheochromocytoma. Pheochromocytoma: recommendations for clinical practice from the First International Symposium. October 2005. Nat Clin Pract Endocrinol Metab. 2007 Feb;3(2):92-102. doi: 10.1038/ncpendmet0396. PMID 17237836
- [Background] Plouin PF, Duclos JM, Soppelsa F, Boublil G, Chatellier G. Factors associated with perioperative morbidity and mortality in patients with pheochromocytoma: analysis of 165 operations at a single center. J Clin Endocrinol Metab. 2001 Apr;86(4):1480-6. doi: 10.1210/jcem.86.4.7392. PMID 11297571
- [Background] Pacak K. Preoperative management of the pheochromocytoma patient. J Clin Endocrinol Metab. 2007 Nov;92(11):4069-79. doi: 10.1210/jc.2007-1720. PMID 17989126
- [Background] Prys-Roberts C, Farndon JR. Efficacy and safety of doxazosin for perioperative management of patients with pheochromocytoma. World J Surg. 2002 Aug;26(8):1037-42. doi: 10.1007/s00268-002-6667-z. Epub 2002 Jun 19. PMID 12192533
- [Background] Bruynzeel H, Feelders RA, Groenland TH, van den Meiracker AH, van Eijck CH, Lange JF, de Herder WW, Kazemier G. Risk Factors for Hemodynamic Instability during Surgery for Pheochromocytoma. J Clin Endocrinol Metab. 2010 Feb;95(2):678-85. doi: 10.1210/jc.2009-1051. Epub 2009 Dec 4. PMID 19965926
- [Background] van der Horst-Schrivers AN, Kerstens MN, Wolffenbuttel BH. Preoperative pharmacological management of phaeochromocytoma. Neth J Med. 2006 Sep;64(8):290-5. PMID 16990692
- [Background] Eisenhofer G, Rivers G, Rosas AL, Quezado Z, Manger WM, Pacak K. Adverse drug reactions in patients with phaeochromocytoma: incidence, prevention and management. Drug Saf. 2007;30(11):1031-62. doi: 10.2165/00002018-200730110-00004. PMID 17973541
- [Background] Kinney MA, Warner ME, vanHeerden JA, Horlocker TT, Young WF Jr, Schroeder DR, Maxson PM, Warner MA. Perianesthetic risks and outcomes of pheochromocytoma and paraganglioma resection. Anesth Analg. 2000 Nov;91(5):1118-23. doi: 10.1097/00000539-200011000-00013. PMID 11049893
- [Background] Eisenhofer G, Bornstein SR. Surgery: Risks of hemodynamic instability in pheochromocytoma. Nat Rev Endocrinol. 2010 Jun;6(6):301-2. doi: 10.1038/nrendo.2010.65. No abstract available. PMID 20502462
- [Background] Karthikeyan G, Moncur RA, Levine O, Heels-Ansdell D, Chan MT, Alonso-Coello P, Yusuf S, Sessler D, Villar JC, Berwanger O, McQueen M, Mathew A, Hill S, Gibson S, Berry C, Yeh HM, Devereaux PJ. Is a pre-operative brain natriuretic peptide or N-terminal pro-B-type natriuretic peptide measurement an independent predictor of adverse cardiovascular outcomes within 30 days of noncardiac surgery? A systematic review and meta-analysis of observational studies. J Am Coll Cardiol. 2009 Oct 20;54(17):1599-606. doi: 10.1016/j.jacc.2009.06.028. PMID 19833258
- [Background] Kim AW, Quiros RM, Maxhimer JB, El-Ganzouri AR, Prinz RA. Outcome of laparoscopic adrenalectomy for pheochromocytomas vs aldosteronomas. Arch Surg. 2004 May;139(5):526-9; discussion 529-31. doi: 10.1001/archsurg.139.5.526. PMID 15136353
- [Background] Shen WT, Grogan R, Vriens M, Clark OH, Duh QY. One hundred two patients with pheochromocytoma treated at a single institution since the introduction of laparoscopic adrenalectomy. Arch Surg. 2010 Sep;145(9):893-7. doi: 10.1001/archsurg.2010.159. PMID 20855761
- [Background] Kocak S, Aydintug S, Canakci N. Alpha blockade in preoperative preparation of patients with pheochromocytomas. Int Surg. 2002 Jul-Sep;87(3):191-4. PMID 12403097
- [Background] Weingarten TN, Cata JP, O'Hara JF, Prybilla DJ, Pike TL, Thompson GB, Grant CS, Warner DO, Bravo E, Sprung J. Comparison of two preoperative medical management strategies for laparoscopic resection of pheochromocytoma. Urology. 2010 Aug;76(2):508.e6-11. doi: 10.1016/j.urology.2010.03.032. Epub 2010 May 23. PMID 20546874
- [Background] Mueller T, Gegenhuber A, Dieplinger B, Poelz W, Haltmayer M. Capability of B-type natriuretic peptide (BNP) and amino-terminal proBNP as indicators of cardiac structural disease in asymptomatic patients with systemic arterial hypertension. Clin Chem. 2005 Dec;51(12):2245-51. doi: 10.1373/clinchem.2005.056648. Epub 2005 Oct 13. PMID 16223888
- [Derived] Buitenwerf E, Osinga TE, Timmers HJLM, Lenders JWM, Feelders RA, Eekhoff EMW, Haak HR, Corssmit EPM, Bisschop PHLT, Valk GD, Veldman RG, Dullaart RPF, Links TP, Voogd MF, Wietasch GJKG, Kerstens MN. Efficacy of alpha-Blockers on Hemodynamic Control during Pheochromocytoma Resection: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2381-91. doi: 10.1210/clinem/dgz188. PMID 31714582